CLINICAL TRIAL: NCT00002018
Title: Double-Blind, Randomized, Dose Ranging Study of Alferon LDO (Low Dose Oral Interferon Alfa-n3 (Human Leukocyte Derived)) in HIV+ Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Interferon Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 069B; 90-355ME
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1993-03

CONDITIONS: HIV Infections
Keywords: Interferon Type I
MeSH Terms: conditions — HIV Infections | interventions — Interferon Alfa-n3

INTERVENTIONS:
Drug: Interferon alfa-n3

SUMMARY:
To conduct a double-blind, randomized, dose ranging study of an orally administered low dose interferon alfa-n3 (IFN-An3) immunomodulator in the treatment of symptomatic HIV+ subjects.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine (AZT).
* Didanosine (ddI)

Patients must have:

* Seropositivity to HIV-1 by ELISA and Western blot.
* At least 1 of the HIV-related clinical symptoms or opportunistic infections listed in protocol.
* Written informed consent.
* If already on zidovudine (AZT) or didanosine (ddI), must have been on this therapy for at least 75 of the 90 days prior to study entry.

Prior Medication:

Allowed:

* Zidovudine (AZT).
* Didanosine (ddI)

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Major active opportunistic infection requiring active care within 2 weeks of study entry.
* Evidence of chronic hepatitis with severe liver dysfunction:
* albumin < 2 g/dl and SGOT or SGPT > 5 x upper limit of normal prothrombin time > 1.5 x upper limit of normal).
* Other active gastrointestinal, renal, respiratory, endocrine, hematologic, cardiovascular, neurologic, or psychiatric disorder.
* Transfusion dependency defined as requiring > 1 unit of packed red blood cells (RBC) per month within 3 months prior to study entry.

Concurrent Medication:

Excluded:

* Experimental medications other than didanosine (ddI).
* Chronic prophylactic use of any topical or systemic fungal medication such as ketoconazole, fluconazole, or clotrimazole.
* Chronic prophylactic use of any topical or systemic anti-viral medication such as acyclovir or ganciclovir except zidovudine (AZT) or didanosine (ddI).

Patients with the following are excluded:

* Asymptomatic at study entry.
* Presence of antibodies to interferon due to prior therapy.
* Hospitalization within 2 weeks of study entry.
* Transfusion dependency.
* Unwilling or unable to give informed consent.
* Evidence of any concurrent organ dysfunction listed in Exclusion Co-Existing Conditions.
* Unlikely or unable to comply with the requirements of the protocol.

Prior Medication:

Excluded within 6 weeks of study entry:

* Interferons.
* Excluded within 45 days of study entry:
* Immunosuppressive agents.
* Chemotherapy.
* Steroids.
* Immunomodulators.
* Isoprinosine.
* BCG vaccine.

Prior Treatment:

Excluded within 2 weeks of study entry:

* Hospitalization.

Active intravenous (IV) drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Med Ctr, New York, New York, United States